CLINICAL TRIAL: NCT05796687
Title: Evaluation of My Future Self, an Innovative Teen Pregnancy Prevention Intervention
Brief Title: Evaluation of My Future Self, an New Teen Pregnancy Prevention Group Intervention for Youth in Non-traditional Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: ETR Associates (Other)
Responsible Party: Principal Investigator, Mona Desai, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHLA-23-00049
Record Dates: First submitted 2023-03-22; First posted 2023-04-03 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Teen Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- My Future Self Intervention (Experimental): My Future Self - 5 group sessions; 1 hour each over 5 weeks; content includes: health education around abstinence and contraception methods, and consideration of goals of parenthood and family planning in their adult future; future plans, discussion of healthy intimate partner relationships/
  Interventions: Behavioral: My Future Self
- Control (No Intervention): Youth will continue to receive any services that they would normally receive around health education.

INTERVENTIONS:
Behavioral: My Future Self — My Future Self is based upon the Theory of Possible Selves, which promotes the capacity of young people to construct goals for a successful adulthood. Youth who hold a balanced set of negative and positive images of their future have both a) a positive goal to strive for and b) awareness of the personally relevant consequences of not meeting that goal. My Future Self also includes two new supportive gaming elements that reinforce learning of relevant knowledge and skills as well as provide opportunities for youth to individually practice these skills in a personalized virtual environment. Gaming interventions using interactive technology can significantly increase self-reported abstinence and lower reports of diagnosed STD in young women, as well as reduce risky sex in high-risk young men who have sex with men. Youth will participate in these gaming elements on tablets provided by CHLA. My Future Self will be implemented as a ninety-minute small group 5-week program.
  Arms: My Future Self Intervention

SUMMARY:
Children's Hospital Los Angeles and ETR will implement and test the effectiveness of a pregnancy prevention intervention, My Future Self, targeting youth ages 16-19 in Los Angeles and San Diego Counties who, for a variety of reasons, are receiving education or training in non-traditional settings. These youth typically experience a combination of needs related to unstable or no housing, extreme poverty, involvement with child welfare or juvenile justice, historical trauma, and/or learning differences. My Future Self is a 5 week program consisting of 5 group sessions. Our study will enroll up to 704 highly mobile youth from various sites in Los Angeles and San Diego. Youth will be randomized to receive the My Future Self intervention in conjunction with their regular services or just their regular services. All youth enrolled will complete baseline, 6 month and 12 month surveys.

DETAILED DESCRIPTION:
Children's Hospital Los Angeles and ETR will implement and test the effectiveness of a pregnancy prevention intervention, My Future Self, targeting youth ages 16-19 in Los Angeles and San Diego Counties who, for a variety of reasons, are receiving education or training in non-traditional settings. These youth typically experience a combination of needs related to unstable or no housing, extreme poverty, involvement with child welfare or juvenile justice, historical trauma, and/or learning differences.

Currently, there are a few evidence-based interventions that focus on sub populations of these youth in alternative schools (All4You!, All4You2!), those at risk for dropping out of school (Crossroads/TCAP), and those coming from out of home care settings (Power Through Choices). However additional interventions are needed as these youth represent a vulnerable population with unique needs and barriers to pregnancy prevention requiring approaches that are tailored to nontraditional educational settings, familial circumstances, developmental trajectory, and that are synergistic with the generational reliance on technology.

ELIGIBILITY:
Inclusion Criteria:

Youth will be eligible for enrollment in the evaluation if they:

* Are served, or identified on outreach, by one of our partner youth-serving agencies or schools
* Are ages 16-19 years
* Are English-language speakers
* Are not currently pregnant
* Have no immediate travel plans (i.e., are planning on being in the area for the length of the intervention)
* Have not previously enrolled in the study, and
* Answer the baseline survey items related to our primary outcome (which will be assessed after completion of the baseline survey).

Exclusion Criteria:

* Outside of age range
* Currently pregnant
* Not planning to be in the area for the length of the intervention)
* Previously enrolled in the study

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 704 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Protection from pregnancy in the past 90 days | Past 90 days
  Had vaginal sex in the past 90 days (% No) OR Used contraception, at least 80% of the time when having vaginal sex (% Yes)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Desai, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No